CLINICAL TRIAL: NCT05037890
Title: The Effects of Plant Sterol and Plant Stanol Ester Enriched Foods on Liver Inflammation in Subjects at Risk to Develop NASH
Brief Title: Effects of Plant Sterols and Stanols on Liver Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Raisio Group (Industry); Unilever R&D (Industry); BASF (Industry)
Responsible Party: Principal Investigator, Jogchem Plat, Professor, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NL70963.068.19
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: Liver inflammation; Plant sterols; Plant stanols
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hepatitis | interventions — Margarine

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double blinded study with a run-period of 2 weeks, an intervention period of 6 months and a wash-out period of 1 month.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Colour-coded margarin tubs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Plant sterol enriched margarine (Active Comparator): 20 grams plant sterol enriched margarine on a daily basis for a period of 6 months.
  Interventions: Dietary Supplement: Margarine
- Plant stanol enriched margarine (Active Comparator): 20 grams plant stanol enriched margarine on a daily basis for a period of 6 months.
  Interventions: Dietary Supplement: Margarine
- Control margarine (Placebo Comparator): 20 grams control margarine on a daily basis for a period of 6 months.
  Interventions: Dietary Supplement: Margarine

INTERVENTIONS:
Dietary Supplement: Margarine — Intake of margarine

SUMMARY:
This study is a randomized, placebo-controlled, double blinded pilot study to assess the effect of consuming plant sterol or plant stanol esters (3 grams/day) for 6 months on ALT concentrations in subjects with elevated ALT concentrations, i.e. who are at risk to develop NASH.

DETAILED DESCRIPTION:
Rationale: As the prevalence of obesity is reaching epidemic proportions, the prevalence of non-alcoholic fatty liver disease (NAFLD), including non-alcoholic steatohepatitis (NASH), increases concomitantly and becomes a major global health hazard. Successful pharmacological interventions to treat or prevent NASH are not available and so far only weight loss has clear benefits, but sustained weight-loss is difficult to achieve on the longer-term. We recently demonstrated in mice that plant sterol and stanol ester consumption inhibited the development of liver inflammation. Moreover, Javanmardi and co-workers recently observed reduced plasma concentrations of Alanine Transaminase (ALT) and Aspartate Transaminase (AST) after daily plant sterol consumption (1.6 g/d) for 6 weeks in a population of adult NAFLD patients. In the current study, we propose to evaluate the effect of long-term consuming plant sterol or plant stanol esters on ALT concentrations in subjects who are at risk to develop NASH. Furthermore, we want to demonstrate the effect of plant sterol and plant stanol consumption on other parameters reflecting liver health, such as cathepsin-D, liver fat and liver insulin sensitivity.

Objective: To assess the effect of consuming plant sterol or plant stanol esters (3 grams/day) for 6 months on ALT concentrations in subjects with elevated ALT concentrations, i.e. who are at risk to develop NASH.

Study design: This study is a randomized, placebo-controlled, double blinded pilot study with a run-period of 2 weeks, an intervention period of 6 months and a wash-out period of 1 month.

Study population: 90 subjects with elevated ALT concentrations (>ULN), aged 18-75 years.

Intervention: All subjects will start a run-in period of two weeks during which they consume daily 20 grams of control margarine after which they will be randomly allocated to consume 20 grams control margarine or plant sterol or plant stanol enriched margarine on a daily basis for a period of 6 months.

Main study parameters/endpoints: The primary outcome parameter in this study is the change in plasma ALT concentration.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: During a screening visit, body weight, body height and blood pressure are determined and a blood sample (5.5 mL) will be drawn. During the run-in period of two weeks, subjects will receive 20g control margarine and during the intervention period of 6 months they will be randomized to receive control, plant sterol ester or plant stanol ester margarine. On 7 occasions a fasting blood sample will be drawn (with a total of 195 mL) and at baseline and in week 26, samples for VOCs analysis will be taken, a FibroScan will be performed to measure liver fat and liver stiffness, body composition will be determined and retinal images will be taken. In a subgroup of 30 subjects, a two-step hyperinsulinemic-euglycemic clamp (278 mL blood sample) including a ventilated hood measurement for indirect calorimetry will be performed and liver fat and liver inflammation will be measured with MRS imaging at baseline and at the of intervention in week 26. All subjects will be asked to fill out a food frequency questionnaire, a physical activity questionnaire and a quality of life questionnaire two times and to keep a diary throughout the study and body weight and blood pressure will be assessed on five occasions.

Venipuncture and insertion of a cannula can cause discomfort and possibly a local haematoma or bruise. Indirect calorimetry might evoke claustrophobic reactions, but there are no physical risks involved. MRS and MRI are modern diagnostic tools that do not imply significant risks (no ionizing radiation). In principle, all measurements are routine in our metabolic research unit (MRUM) and are not expected to lead to physical side effects. Total time investment spread-out over the study participation will be approximately 7 hours or 34 hours (depending on the subgroup), excluding travel time. Plant sterol and plant stanol enriched products are commercially available and we therefore do not foresee any risks related to the consumption of these food products

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent
2. Elevated ALT concentrations (>50 U/L for men and >40 U/L for women)
3. Metabolic syndrome according to the NCEP ATP III definition (Grundy 2005)
4. Aged between 18 and 75 years
5. Willingness to consume 20 grams of margarine provided by us on a daily basis for a period of 6 months

Exclusion Criteria:

1. Are less than 18 years of age or over 75 years of age
2. Females who are pregnant, breast feeding or who may wish to become pregnant during the study
3. Have a significant acute or chronic coexisting illness such as cardiovascular disease, chronic kidney disease, gastrointestinal disorder, endocrinological disorder, immunological disorder, cancer or any condition which contraindicates, in the investigator's judgement, entry to the study
4. Severe medical conditions that might interfere with the study such as epilepsy, asthma, chronic obstructive pulmonary disease, inflammatory bowel disease and rheumatoid arthritis
5. Use of diuretics or insulin therapy
6. History of illicit drug use
7. Consume more than the recommended alcohol guidelines i.e. >21 alcohol units/week for males and >14 units/week for females
8. Not willing to stop the consumption of plant sterol or plant stanol enriched products 1 month before the start of the study (wash-in period)
9. Use of an investigational product in another biomedical study within the previous month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Liver inflammation | 6 months
  ALT levels

SECONDARY OUTCOMES:
Glucose metabolism | 6 months
  Insulin sensitivity using a 2-step clamp

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No